CLINICAL TRIAL: NCT00006682
Title: An Open-Label Phase II Study of Navelbine (Vinorelbine Tartrate) and Taxotere (Docetaxel) as First-Line Therapy for Metastatic Breast Cancer
Brief Title: Vinorelbine and Docetaxel in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068284; WHC-2000056; NCI-V00-1631
Record Dates: First submitted 2000-12-06; First posted 2004-05-04 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2001-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Vinorelbine

STUDY DESIGN:
Intervention Model Description: Open-Label Navelbine (vinorelbine tartrate) and Taxotere (docetaxel) as First-Line Therapy for Metastatic Breast Cancer
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel — Docetaxel 70mg/m2 on day 1 of every 21-day cycle
  Other Names: Taxotere
Drug: vinorelbine ditartrate — Navelbine 20mg/m2 on Day 1 and D8 of a 21-day cycle
  Other Names: Navelbine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vinorelbine combined with docetaxel in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate in women with metastatic breast cancer treated with vinorelbine and docetaxel. II. Determine the time to disease progression, time to treatment failure, response duration, and survival in this patient population treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive vinorelbine IV on days 1 and 8, and docetaxel IV over 1 hour on day 1 only. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed for 1 month, and then every 1.5-3 months for 1 year.

PROJECTED ACCRUAL: Approximately 69 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IV breast cancer Disease progression following prior adjuvant chemotherapy (no disease progression during treatment with prior doxorubicin) Bidimensionally measurable disease Prior radiotherapy allowed if disease completely outside radiation port or histologic evidence of measured area indicating malignancy and not radiation fibrosis No CNS metastases Brain metastases previously treated with radiotherapy or surgical excision allowed if no evidence of residual metastases on brain CT or MRI Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Over 18 Sex: Female Menopausal status: Premenopausal or postmenopausal Performance status: ECOG 0-1 Life expectancy: Greater than 16 weeks Hematopoietic: WBC at least 2,000/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin less than 2.0 mg/dL SGOT/SGPT less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase less than 2.5 times ULN Renal: Not specified Cardiovascular: No symptomatic New York Heart Association class II or greater congestive heart failure No significant arrhythmia requiring drug therapy No myocardial infarction within the past 6 months No uncontrolled cardiac disease or unstable angina Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix No preexisting clinically significant peripheral neuropathy (no prior neuropathy of any grade if previously treated with paclitaxel) No unstable, preexisting medical condition No serious active infection No other underlying medical, psychological, familial, sociologic, or geographic condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 7 days since prior hematopoietic growth factors (filgrastim (G-CSF), sargramostim (GM-CSF), or epoetin alfa) At least 7 days since prior platelet transfusion Chemotherapy: See Disease Characteristics No prior vinca alkaloids (including vinorelbine or docetaxel) No other concurrent antineoplastic agents Endocrine therapy: No concurrent anticancer hormonal agents Radiotherapy: See Disease Characteristics No concurrent palliative radiotherapy Surgery: See Disease Characteristics Other: No other concurrent investigational drug or device

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2002-01-22 (Actual); Study Completion 2002-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Perry, MD, Study Chair — Medstar Health Research Institute
Locations (2):
- United States (2):
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia